CLINICAL TRIAL: NCT01043432
Title: Executive Dysfunction and Suicide in Psychiatric Outpatients and Inpatients
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: D7210-R
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Traumatic Brain Injury; Suicidality
Keywords: Traumatic Brain Injury; Suicide; Executive Function
MeSH Terms: conditions — Brain Injuries, Traumatic; Suicidal Ideation; Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Moderate/severe TBI and history of suicidal behavior Group 1: Moderate/severe TBI and history of suicidal behavior
- Moderate/Severe TBI and no history of suicidal behaviorGroup: Moderate/Severe TBI and no history of suicidal behavior
- No TBI and a history of suicidal behavior Group 3: No TBI and a history of suicidal behavior
- No TBI and no history of suicidal behavior Group 4: No TBI and no history of suicidal behavior

SUMMARY:
Those with traumatic brain injury (TBI) are at increased risk for suicidal behavior, and suicidality is associated with executive dysfunction. In the aim of highlighting an important risk factor, this study will assess decision making in the context of an interaction between suicide and TBI. Findings will also allow for exploratory analyses aimed at identifying associations between performance on measures of executive functioning and psychological distress. The long-term objective of this study is to increase understanding regarding executive dysfunction, as a multidimensional construct, with the ultimate goal of conceptualizing assessment tools and interventions aimed at decreasing suicidality in the at-risk population of veterans with a history of TBI.

DETAILED DESCRIPTION:
Recent studies indicate that veterans who engage in suicidal behavior have a history of traumatic brain injury (TBI), and veterans with a history of TBI engage in suicidal behavior. Existing research also suggests an association between suicidality and executive dysfunction (e.g., impaired decision making). To date a clearly defined study has not been conducted to explore the relationship between executive dysfunction as a multidimensional construct (i.e., decision making, impulsivity, concept formation, and aggression) and suicidal behavior in the vulnerable population of those with a history of moderate to severe TBI. Increased understanding regarding this at-risk population is necessary to facilitate the creation of appropriate assessment strategies and interventions. This study will assess decision making in the context of an interaction between suicide and TBI. Findings will also allow for exploratory analyses aimed at identifying associations between performance on measures of executive functioning and psychological distress. Toward this end, the present study seeks to compare test performance among four well-defined groups of veterans: (1) those with moderate to severe TBI and a history of suicidal behavior; (2) those with moderate to severe TBI and no history of suicidal behavior; (3) those with no TBI and a history of suicidal behavior; (4) and those with no TBI and no history of suicidal behavior. This grant proposal is in direct support of the Rehabilitation Research and Development goal of maximizing functional recovery in those with TBI by potentially: 1) increasing clinicians' ability to identify neuropsychological correlates of suicidal behavior for those with moderate to severe TBI; 2) identifying psychometrically sound measures of executive functioning that correspond to real-life behaviors that impact treatment response and recovery; 3) facilitating the creation of innovative assessment techniques and psychosocial interventions (e.g., safety planning) to minimize complications in the management of suicidal behavior due to TBI-related impairments; and 4) creating a basis for further and much-needed research in this area. Ultimately, findings from this study would both contribute to clinicians' ability to identify veterans with TBI who are at risk for suicidal behavior, and create a foundation on which to base further research regarding the relationships between cognition, emotional distress, and suicidality in TBI survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* Ability to provide adequate effort (CARB score of Type 1 or 2)
* Determination of positive or negative history of moderate or severe TBI
* Determination of positive or negative history of suicidal behavior
* Ability to adequately respond to questions regarding the informed consent procedure

Exclusion Criteria:

* Diagnosis of neurological conditions other than moderate or severe TBI
* Inability to adequately respond to questions regarding the informed consent procedure
* Inability to provide adequate effort (CARB score of Type 3 or 4)
* History of a psychotic or bipolar I mood disorder
* History of drug or alcohol abuse in the past 7 days
* Participating in another study in which the results of this study may be impacted
* History of non-alcohol substance abuse within the last 30 days as identified on the SCID substance use module
* History of same-day drug or alcohol abuse as identified on the UWRAP pre-administration questionnaire Veterans who report using substances the day of the study visit will be placed on hold and will be rescreened in 30 and 60 days
* History of mild TBI only

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants in this observational study will be all individuals willing and eligible from the following populations: 1) those admitted to the locked inpatient psychiatric unit at the Eastern Colorado Health Care System (ECHCS) Denver VA Medical Center (VAMC); 2) those seeking outpatient mental health, rehabilitative, or psychological or other services at the Denver VAMC or Colorado Springs Community Based Outpatient Clinic (CBOC) or other CBOC's; 3) those in an ECHCS domiciliary (e.g., Valor Point); 4) those on existing clinical and research databases; and 5) veterans in the community not seeking care within the Veterans Health Administration (VHA).
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2010-06; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Anne Brenner, PhD, Principal Investigator — VA Eastern Colorado Health Care System, Denver
Locations (1):
- VA Eastern Colorado Health Care System, Denver, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Moderate/severe TBI and history of suicidal behavior = 22
- Group 2: Moderate/Severe TBI and no history of suicidal behavior = 51
- Group 3: No TBI and a history of suicidal behavior = 12
- Group 4: No TBI and no history of suicidal behavior = 48
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 22 | 51 | 12 | 48
Completed | 22 | 51 | 12 | 48
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Moderate/Severe TBI and no History of Suicidal behaviorGroup 2: Moderate/Severe TBI and no history of suicidal behavior
- Total: Total of all reporting groups
Arm/Group | Moderate/Severe TBI and History of Suicidal Behavior Group 1 | Moderate/Severe TBI and no History of Suicidal behaviorGroup 2 | No TBI and a History of Suicidal Behavior Group 3 | No TBI and no History of Suicidal Behavior Group 4 | Total
Number analyzed (Participants) | 22 | 51 | 12 | 48 | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 51 | 12 | 48 | 133
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (10.3) | 53 (8.5) | 51.7 (12) | 54.2 (7.6) | 52.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 4 | 8 | 15
  Male | 19 | 51 | 8 | 40 | 118
Region of Enrollment [Number; unit: participants]
  United States | 22 | 51 | 12 | 48 | 133
History of TBI (Present or Absent) - Lifetime OSU TBI-ID [Number; unit: participants] — Lifetime History TBI (Present or Absent)
  participants | 22 | 51 | 0 | 0 | 73

OUTCOME MEASURES:

1. Primary Outcome: Iowa Gambling Test
Description: Iowa Gambling Test - Total Raw Score The Iowa Gambling task requires examinees to sit in front of a computer screen displaying four decks of cards (Decks A, B, C, and D) and select a card from any of the four decks. Decks A and B are the disadvantageous decks because they produce high immediate gains however over time examinees will experience a higher loss. Decks C and D are the advantageous decks because they produce lower gains but over time examinees will experience smaller losses. Examinees will make 100 choices (trials). To measure performance, the 100 trials are divided, in order, into 5 'blocks' of 20. A net score is calculated for each block as the number of cards selected from the advantageous decks minus the disadvantageous decks and the total raw score is the sum of the scores for blocks 1-5. The overall total score can range from -100 (worst outcome) to 100 (best outcome)and the score for each block can range from -20 to 20
Time Frame: One time - for the vast majority of participants the research protocol was initiated directly after informed consent procedures were completed (within hours). Negative values are possible with this measure, see Outcome Description.
Measure: Mean (Standard Deviation); unit: Total Raw on a scale from -100 to 100
Groups:
- Group 1: Moderate/severe TBI and history of suicidal behavior
- Group 2: Moderate/Severe TBI and no history of suicidal behavior
- Group 3: No TBI and a history of suicidal behavior
- Group 4: No TBI and no history of suicidal behavior
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 22 | 50 | 12 | 48
Total Raw on a scale from -100 to 100 | -4.2 (27.7) | 1.7 (26.6) | 3.5 (24.5) | 5.3 (25.5)
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3 vs Group 4; Linear regressions were utilized to model the outcomes of interest as a function of SA, TBI group, and the interaction between the two groups; Test type: Superiority or Other; p > .05, Regression, Linear

ADVERSE EVENTS:
Arm/Group | All Groups
Serious Adverse Events (participants affected / at risk) | 0/133
Other Adverse Events (participants affected / at risk) | 0/133

LIMITATIONS AND CAVEATS:
Majority of control group had lifetime history of psychiatric disorders Significant challenges with recruiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes